CLINICAL TRIAL: NCT04483297
Title: First-In-Human Study of AK1320 Encapsulated Microspheres (AK1320 MS) In Subjects With Degenerative Spondylolisthesis and Concomitant Symptomatic Spinal Stenosis Who Are Undergoing Decompression And Single Level Instrumented Posterolateral Lumbar Autograft Fusion Surgery
Brief Title: First-In-Human Study of AK1320 Encapsulated Microspheres (AK1320 MS)
Acronym: ENHANCE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Asahi Kasei Pharma Corporation (Industry)
Collaborators: Emergent Clinical Consulting, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK1320-101
Record Dates: First submitted 2020-07-14; First posted 2020-07-23 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Degenerative Spondylolisthesis; Spinal Stenosis
Keywords: degenerative spondylolisthesis; spinal stenosis; posterolateral lumber fusion surgery; autograft
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK1320 MS (Experimental): AK1320 MS + Local Autologous Bone + Posterior Fixation
  Interventions: Drug: AK1320 MS
- Control (Other): Local Autologous Bone + Posterior Fixation
  Interventions: Other: Control

INTERVENTIONS:
Drug: AK1320 MS — AK1320 MS + Local Autologous Bone + Posterior Fixation. Ascending Dose.
  Arms: AK1320 MS
Other: Control — Local Autologous Bone + Posterior Fixation
  Arms: Control

SUMMARY:
The safety and efficacy of AK1320 MS will be evaluated in patients with degenerative spondylolisthesis and concomitant symptomatic spinal stenosis who are undergoing decompression and single level instrumented posterolateral lumber autograft fusion surgery.

DETAILED DESCRIPTION:
This will be a first in human Phase I, ascending dose, multi-center, randomized patient study evaluating the efficacy, safety, PK of AK1320 MS. The study will enroll up to 4 dose escalating cohorts with each cohort having 2 treatment groups. Cohort 1 and Cohort 2 (AK1320 MS group (n=3-7); Control group (n=0-3)) and Cohort 3 and Cohort 4 (AK1320 MS group (n=6-7); Control group (n=0-3)).

ELIGIBILITY:
Inclusion Criteria:

1. Involved level L1 to S1
2. Use of local autologous bone only.
3. Degenerative spondylolisthesis up to Meyerding's Classification Grade 1 or 2.
4. Moderate or higher disability as assessed by Oswestry Disability Index.
5. Neurogenic claudication and/or radiculopathy with or without back pain.
6. Male or female over 22 years of age and less than 81 years of age.

Exclusion Criteria:

1. Prior lumbar decompression or spine fusion attempt (any level).
2. Undergoing concurrent interbody fusion.
3. Requires spinal fusion at more than one lumbar level.
4. Degenerative scoliosis.
5. BMI > 40.
6. Radiographically confirmed significant spinal instability.
7. Active or recent (within the past two (2) years) worker's compensation litigation.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events | 24 months
Summary of Neurological Status | 24 months
  Neurological status will be determined preoperatively and postoperatively using a comprehensive neurological status scale. Neurological status is based on four types of measurements: lower extremity motor, dermatomal sensation, reflexes and straight leg raise.

SECONDARY OUTCOMES:
Successful Fusion | 24 months
  Fusion will be evaluated through CT scans. Successful fusion will be defined as complete bridging bone between the index level transverse processes with a lack of lucency or lucent lines through the fusion mass.
Oswestry Low Back Pain Disability Questionnaire (ODI) | 24 months
36-Item Short Form Survey (SF-36v2®) | 24 months
AK1320 plasma concentrations | Pre-op(day 0), Post-op (day 0, day1), 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks and 6 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (7):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal General Hospital, Montreal, Quebec
  - Hôpital Sacré-Coeur de Montréal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Québec Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No